CLINICAL TRIAL: NCT02614014
Title: Effect of the Stress and Personality Profiles in the Development, Evolution and Treatment of Inflammatory Bowel Disease.
Brief Title: Stress and Personality Profiles in IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asociación Española de Gastroenterología (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSI-EII-09
Record Dates: First submitted 2015-09-28; First posted 2015-11-25 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

ARMS (2):
- Psychological intervention (Experimental): Cognitive-behavior interventional program
  Interventions: Behavioral: Cognitive-behavior interventional program
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Cognitive-behavior interventional program
  Arms: Psychological intervention

SUMMARY:
Main aim is to evaluate the role of stress in the evolution of inflammatory bowel disease (IBD) and the quality of life of these patients. A second aim is to establish the existence of any psicopathological profile in these patients. We designed a prospective experimental study were patients are randomized to receive or not a cognitive-behavior program. Patients will be evaluated at 3 and 12 months after the program and study variables will be measured: stress level, coping strategies, quality of life, activity of disease and biological variables related to IBD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years
* Informed consent
* Crohn's disease or ulcerative colitis diagnosis
* Active disease in the last 18 months

Exclusion Criteria:

* Severe mental disease
* Other severe concomitant disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in IBD activity at short and long-term | Measured at baseline, and evaluation at short-term (3 months) and long-term 12 months
  Number of clinical episodes of activity of IBD
Change in IBD activity at short and long-term | Measured at baseline, and evaluation at short-term (3 months) and long-term 12 months
  Number of hospital admisions because of IBD
Change in IBD activity at short and long-term | Measured at baseline, and evaluation at short-term (3 months) and long-term 12 months
  Activity index vaules (CDAI for Crohn's disease and Mayo score for ulcerative colitis)

SECONDARY OUTCOMES:
Change in stress scales at short and long-term | Measured at baseline, and evaluation at short-term (3 months) and long-term 12 months
  Perceived Stress Scale (PSS)
Change in quality of life at short and long-term | Measured at baseline, and evaluation at short-term (3 months) and long-term 12 months
  Inflammatory bowel disease quality-of-life scale (IBDQ)
Change in anxiety and depression at short and long-term | Measured at baseline, and evaluation at short-term (3 months) and long-term 12 months
  HAD scale
Change in stress scales at short and long-term | Measured at baseline, and evaluation at short-term (3 months) and long-term 12 months
  Disease related stress scale (EAE)
Change in stress scales at short and long-term | Measured at baseline, and evaluation at short-term (3 months) and long-term 12 months
  Vital stressors scale (AVE)
Change in stress scales at short and long-term | Measured at baseline, and evaluation at short-term (3 months) and long-term 12 months
  stress coping questionnaire (CAE)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Van der Hofstadt, Study Director — Hospital General Universitario de Alicante
Locations (1):
- Department of health psychology. Hospital General Universitario de Alicante, Alicante, Spain

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Bernabeu P, van-der Hofstadt C, Rodriguez-Marin J, Gutierrez A, Alonso MR, Zapater P, Jover R, Sempere L. Effectiveness of a Multicomponent Group Psychological Intervention Program in Patients with Inflammatory Bowel Disease: A Randomized Trial. Int J Environ Res Public Health. 2021 May 19;18(10):5439. doi: 10.3390/ijerph18105439. PMID 34069621